CLINICAL TRIAL: NCT02981563
Title: Time Together: A Multi-site Nursing Intervention Project Using a Single System Experimental Design
Acronym: TT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 350000210
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-11

CONDITIONS: Mental Health Nursing; Nurse-Patient Relations
Keywords: engagement; psychiatric in-patient care; mental health nursing; quality interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Time Together (Experimental): Time Together as described under "Interventions"
  Interventions: Other: Time Together

INTERVENTIONS:
Other: Time Together — For a fixed time during the day, staff dedicates their time to exclusively engage with the patients. Different activities will be offered to both patients and staff, such as playing board games, taking a walk, or having individual conversations. Other duties of more administrative nature, visits and meetings will be performed at other times during the day. Through this, opportunities for interaction are both created and protected.
  Other Names: Protected Engagement Time

SUMMARY:
The aim of this project is to test and evaluate a nursing intervention, Time Together (TT), created to enable quality interactions between patients and staff in psychiatric inpatient care. The research questions are:

Does TT influence the quality of interactions between staff and patients? Does TT influence patients' levels of anxiety and depressive symptoms? Does TT influence staffs' levels of perceived stress and levels of stress of conscience? Does TT influence the prevalence of coercive measures, mean length of hospital stay and the use of PRN medication?

In parallel, a process evaluation will be conducted, answering questions such as:

How do staff and patients describe their experiences of the intervention and how do contextual factors influence the effects of the intervention? What are the relationship between the outcome variables and the degree of compliance with the intended intervention? What problems are there with recruitment and dropouts?

DETAILED DESCRIPTION:
BACKGROUND:

Despite the long known significance of the nurse-patient relationship, research in psychiatric inpatient care still reports on unfulfilled expectations of, and difficulties in interactions and relationships between patients and staff. As one solution to the contemporary circumstances, interventions that creates structures that allow quality interactions between patients and staff are needed.

INTERVENTION TT is an intervention, developed from the intervention Protected Engagement Time. The structure of TT is that staff, for a fixed time during the day, dedicates their time to exclusively engage with the patients. Other duties of more administrative nature, visits and meetings are organized to be performed at other times during the day. This structure will be tested at three psychiatric inpatient care wards in the north of Sweden.

DESIGN AND METHODS An experimental single system design (A-B-Follow-up) will be used. As TT will be introduced as a routine ward activity during the B phase, all patients and staff on the participating wards will be participating in TT. However, participating in the evaluation will be voluntary. Data will be collected through questionnaires once every seventh weekday during 5 weeks for the A phase, and 12 weeks during B phase.

In parallel, a process evaluation will be conducted using semi structured interviews and participating observations.

ELIGIBILITY:
Inclusion criteria for patients:

* 18 years or older
* Admitted to the wards during either A phase, B phase and/or follow-up
* Experience of at least one TT session is required to participate in the B phase

Exclusion criteria for patients:

- Does not master the Swedish language well enough to complete questionnaires and participate in interviews.

Inclusion criteria for staff:

- Regularly employed at the ward during A and B phase and/or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Quality of interactions [patients] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  This is measured using The Caring Professional Scale (CPS) that consists of 14 items answered on a 5-point Likert scale.
Perceived stress [staff] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  PSS consists of 10 items answered on a 5-point Likert scale

SECONDARY OUTCOMES:
Global quality of interactions [patients, staff] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  A 100 mm Visual Analogue Scale expressing the most positive and the most negative rating will be anchored at each end
Anxiety and depressive symptoms [patients] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  The Hospital Anxiety and Depression Scale (HAD) will be used to measure anxiety and depressive symptoms. All items are scored on a 4-point scale.
Stress of Conscience [staff] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  The Stress of Conscience Questionnaire (SCQ) will be used to measure the frequencies of stressful situations and the degree to which these lead to stress of conscience among staff.
Quality of care [staff] | Changes during baseline and intervention period (measured every seventh week day for a total of 16 weeks)
  The Quality in Psychiatric Care- Inpatient Staff (QPC-IPS) questionnaire will be used to measure quality of care.
Number of PRN medications given | Changes during baseline and intervention period (measured weekly for a total of 16 weeks)
  Data will be retrieved from ward registers.
Length of hospital stay | Changes during baseline and intervention period (measured weekly for a total of 16 weeks)
  Data will be retrieved from ward registers.
Use of coercion and violent situations | Changes during baseline and intervention period (measured weekly for a total of 16 weeks)
  Data will be retrieved from ward registers.

REFERENCES:
- [Derived] Molin J, Lindgren BM, Graneheim UH, Ringner A. Does 'Time Together' increase quality of interaction and decrease stress? A study protocol of a multisite nursing intervention in psychiatric inpatient care, using a mixed method approach. BMJ Open. 2017 Aug 28;7(8):e015677. doi: 10.1136/bmjopen-2016-015677. PMID 28851774